CLINICAL TRIAL: NCT05621538
Title: A Combined Neurofeedback-TMS Intervention for Alcohol Use Disorder
Acronym: CNT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Samantha Fede, Assistant Professor, Auburn University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 22145; R00AA027830 (NIH)
Record Dates: First submitted 2022-10-26; First posted 2022-11-18 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder
Keywords: treatment seeking; alcohol; TMS; neurofeedback; supplemental intervention; heavy drinking; problems with drinking
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The PI will prospectively assign treatment groups with blind codes and so will not be blind to treatment type. Other staff, who are the individuals primarily working with the patients and who will be conducting follow-up interviews, will be blind to treatment type. It is not possible to blind the 5th condition (treatment as usual with a brief check-in).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Neurofeedback-active + TMS-active (Experimental): 4 sessions of: TMS (protocol: 10 Hz pulses delivered at 110% of MT in 60 x 5 sec trains with 25 sec ITI) Neurofeedback (protocol: presentation of own brain activity from multiple ROIs measured using fMRI)
  Interventions: Behavioral: Realtime fMRI Neurofeedback - Active; Device: TMS - Active
- Neurofeedback-active + TMS-sham (Active Comparator): 4 sessions of: TMS (protocol: 10 Hz pulses delivered using the Sham TMS coil in 60 x 5 sec trains with 25 sec ITI) Neurofeedback (protocol: presentation of own brain activity from multiple ROIs measured using fMRI)
  Interventions: Behavioral: Realtime fMRI Neurofeedback - Active; Device: TMS - Sham
- Neurofeedback-sham + TMS-active (Active Comparator): 4 sessions of: TMS (protocol: 10 Hz pulses delivered at 110% of MT in 60 x 5 sec trains with 25 sec ITI) Neurofeedback (protocol: presentation of other's brain activity from multiple ROIs measured using fMRI)
  Interventions: Device: TMS - Active; Behavioral: Realtime fMRI Neurofeedback - Yoked Sham
- Neurofeedback-sham + TMS-sham (Sham Comparator): 4 sessions of: TMS (protocol: 10 Hz pulses delivered using the Sham TMS coil in 60 x 5 sec trains with 25 sec ITI) Neurofeedback (protocol: presentation of other's brain activity from multiple ROIs measured using fMRI)
  Interventions: Behavioral: Realtime fMRI Neurofeedback - Yoked Sham; Device: TMS - Sham
- Check-In Only (No Intervention): 4 sessions of: Completing typical pre-TMS/MRI procedures Being prompted to reflect on outside treatment (TAU)

INTERVENTIONS:
Behavioral: Realtime fMRI Neurofeedback - Active — fMRI aided reinforcement of craving regulation
  Arms: Neurofeedback-active + TMS-active; Neurofeedback-active + TMS-sham
Device: TMS - Active — rTMS to right dorsolateral prefrontal cortex to reduce craving
  Other Names: Magventure Magpro
  Arms: Neurofeedback-active + TMS-active; Neurofeedback-sham + TMS-active
Behavioral: Realtime fMRI Neurofeedback - Yoked Sham — Display of feedback from other participant's sessions to serve as a sham for fMRI aided reinforcement of craving regulation
  Arms: Neurofeedback-sham + TMS-active; Neurofeedback-sham + TMS-sham
Device: TMS - Sham — rTMS using placebo coil (no brain stimulation, emulates other features of active TMS), placed over right dorsolateral prefrontal cortex
  Arms: Neurofeedback-active + TMS-sham; Neurofeedback-sham + TMS-sham

SUMMARY:
The goal of this clinical study is to test the effectiveness of a supplemental fMRI neurofeedback and/or TMS intervention in individuals seeking treatment for Alcohol Use Disorder.

After an initial visit, participants will come in once a week for four (4) weeks for an intervention session, which may or may not include TMS and MRI. Participants will be contacted for monthly follow-ups (remotely) for up to 12 months and will be asked to come in for two MRI follow-ups at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19-65
2. Receiving treatment for Alcohol Use Disorder

Exclusion Criteria:

1. MRI Contraindications

   1. Presence of metal in the body that would make having a 7T MRI unsafe (including facial tattoos)
   2. Claustrophobia, such that individual would be unable to stay in the MRI for up to 1 hr
   3. Hearing loss, including tinnitus, that might be made worse by MRI or TMS
2. TMS Contraindications

   1. Has ever had a seizure, or has a family history of epilepsy
   2. Taking medications or substances that lower the seizure threshold
   3. Implanted devices that are in the head or rely on physiological signals
   4. History of neurological disease, such as stroke or brain tumor
   5. Head injury with loss of consciousness greater than 30 minutes
   6. Actively withdrawing from alcohol
3. Family history of schizophrenia or presence of psychotic symptoms

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol Use over Time | Assessed at weeks: 1 (baseline), 2-5 (intervention sessions, pre and post), 9, 13, 17, 21, 25, 33, 37, 41, 45, 49, 53 (follow-ups)
  Alcohol Timeline Followback (alc-TLFB)
Change in Alcohol Craving over Time | Assessed at weeks: 1 (baseline), 2-5 (intervention sessions, pre and post), 9, 13, 17, 21, 25, 33, 37, 41, 45, 49, 53 (follow-ups)
  Alcohol Craving Questionnaire (ACQ)
Change in Community Functioning over Time | Assessed at weeks: 1 (baseline), 2-5 (intervention sessions), 9, 13, 17, 21, 25, 33, 37, 41, 45, 49, 53 (follow-ups)
  Drinker Inventory of Consequences (DrInC)
Change in Employment Status over Time | Assessed at weeks: 1 (baseline), 2-5 (intervention sessions), 9, 13, 17, 21, 25, 33, 37, 41, 45, 49, 53 (follow-ups)
  self-reported employment status
Change in Aggression and Victimization over Time | Assessed at weeks: 1 (baseline), 2-5 (intervention sessions), 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 53, 57 (follow-ups)
  Revised Conflict Tactics Scales (CTS-R)
Change in Antisocial Behavior over Time | Assessed at weeks: 1 (baseline), 2-5 (intervention sessions), 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 53, 57 (follow-ups)
  number of self-reported contacts with the police, convictions, and other criminal behaviors
Change in Brain Activity during Alcohol Cue Presentation over Time | Assessed at weeks: 1 (baseline), 5 (post final intervention), 29 and 57 (follow-ups)
  Measured via fMRI; standard alcohol cue reactivity
Change in Brain Activity during Simultaneous Sociomoral & Alcohol Cue Presentation over Time | Assessed at weeks: 1 (baseline), 5 (post final intervention), 29 and 57 (follow-ups)
  Measured via fMRI; alcohol-cued sociomoral processing

SECONDARY OUTCOMES:
Change in Brain Gray Matter Structure over Time | Weeks: 1 (baseline), 5 (post final intervention), 29 and 57 (follow-ups)
  Measured via MRI; gray matter volume
Change in Brain White Matter Structure over Time | Weeks: 1 (baseline), 5 (post final intervention), 29 and 57 (follow-ups)
  Measured via MRI; white matter diffusion
Change in Resting State Functional Connectivity over Time | Weeks: 1 (baseline), 5 (post final intervention), 29 and 57 (follow-ups)
  Measured via fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Samantha J Fede, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared within the NIAAA Data Archive according to the standard data sharing plan. Deidentified individual data regarding the outcome variables (clinical and MRI) will be included. Participants will have the option to opt out of sharing their individual data.
  Given the highly sensitive and confidential nature of the information, and the magnitude of potential harms to participants associated with disclosure, clinical outcome data pertaining to criminal acts and illegal activities will not be available in the data repository.